CLINICAL TRIAL: NCT00508872
Title: Single-Institution Phase II Trial of Oxaliplatin, 5-Fluorouracil, Leucovorin and Bevacizumab (Folfox-B) for Initially Unresectable Colorectal Liver Metastases: Downstaging Followed By Hepatic Resection
Brief Title: Folfox-B Study for Patients With Colorectal Liver Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual, study terminated.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0816
Record Dates: First submitted 2007-07-27; First posted 2007-07-30 (Estimated); Results first posted 2010-11-04 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Colorectal Liver Metastases
Keywords: Colorectal Liver Metastases; Oxaliplatin; Eloxatin; Fluorouracil; Leucovorin; Bevacizumab; Anti-VEGF monoclonal antibody; rhuMAb-VEGF; Folfox-B; 5-FU; Avastin
MeSH Terms: interventions — Fluorouracil; Bevacizumab; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FOLFOX-B (Experimental): FOLFOX-B: 5-Fluorouracil 400 mg/m^2 IV + Bevacizumab 5 mg/kg IV + Leucovorin 400 mg/m^2 IV + Oxaliplatin 85 mg/m^2 IV
  Interventions: Drug: 5-Fluorouracil; Drug: Bevacizumab; Drug: Leucovorin; Drug: Oxaliplatin

INTERVENTIONS:
Drug: 5-Fluorouracil — 400 mg/m^2 IV over 15 minutes, followed by 2400 mg/m^2 IV Over 46 Hours
  Other Names: 5-FU; Adrucil; Efudex
Drug: Bevacizumab — 5 mg/kg IV Over 30-90 Minutes On Day 1 Every 14 Days
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
Drug: Leucovorin — 400 mg/m^2 IV Over 2 Hours On Day 1 Every 14 Days
  Other Names: Citrovorum; Wellcovorin
Drug: Oxaliplatin — 85 mg/m^2 IV Over 2 Hours On Day 1 Every 14 Days
  Other Names: Eloxatin

SUMMARY:
Objective:

* To evaluate the efficacy of the use of the combination of oxaliplatin, 5-fluorouracil, leucovorin and bevacizumab (FOLFOX-B) in patients with unresectable colorectal liver metastases, with the objective to downstage hepatic disease and enable complete resection of residual disease.

Primary Objective:

* To evaluate the resection rate in patients with initially unresectable hepatic colorectal metastases downstaged with FOLFOX-B. Complete resection of all liver lesions is the goal.

Secondary Objectives:

* To evaluate the probability of complete response, partial response or stable disease.
* To evaluate the proportion of patients who are resected, and the proportion of patients achieving an R0 resection (among those receiving surgery).
* To correlate survival with downstaging and resection based on metastatic colorectal prognostic score.
* To evaluate the disease-free survival and overall survival.
* To evaluate the positron emission tomography response rate.
* To explore correlations of clinical response with telomerase and hTERT expression.

DETAILED DESCRIPTION:
Oxaliplatin and bevacizumab are chemotherapy drugs that are designed to kill cancer cells. 5-FU is a chemotherapy drug that helps to stop the growth of cancer cells. Leucovorin is a drug that may help increase the effect of 5-FU.

The study drugs will be given to you on an outpatient basis and will involve a minimum of 4 cycles and up to a maximum of 12 cycles of chemotherapy. All chemotherapy will be given through a catheter placed in a vein in the shoulder in "cycles". Each "cycle" equals 14 days. On the first day (Day 1) of each cycle, bevacizumab will be given for 30 to 90 minutes and oxaliplatin and leucovorin for 2 hours. On Day 1 as well, part of the total 5-FU dose will be given for 15 minutes through the catheter. The rest of the 5-FU dose is then given through a pump over the next 46 hours. After 46 hours, you will have a rest period, without drug treatment for the rest of the cycle until the start of the next cycle.

Before each chemotherapy cycle, you will have blood drawn (about 2 tablespoons) for tests to check for any side effects. Depending on the results of the blood tests, these blood tests may be done more often. You will also have your vital signs (blood pressure, breathing, temperature, and heart rate) monitored during the treatment. You will be seen every 2 weeks by one of your doctors during your therapy.

If at any time the disease gets worse or you experience any intolerable side effects, you will be taken off the study.

After completion of the 4th cycle of chemotherapy, you will have a complete physical exam and routine blood tests (about 2 tablespoons). You will also have a CT scan of the abdomen and pelvis and a chest x-ray or CT scan of the chest. These tests are being done to find out if the tumor can be removed by surgery.

If your tumors cannot be removed at this time, you will continue to receive the same dose of chemotherapy with the same tests for up to a maximum of 12 cycles. If it is found that the tumor still cannot be removed after 12 cycles, your participation in this study will be complete and your doctor will discuss other treatment options with you.

If the tumor can be removed, you will receive 1 additional cycle of oxaliplatin, leucovorin, and 5-FU (no bevacizumab) at the same doses before you go on to have the surgery. Your surgery will be scheduled 8-12 weeks after the completion of chemotherapy. The surgeon will explain the surgery and any risks. During liver tumor surgery, normal tissue around the edges of the tumor will be collected as part of routine care. You will be asked to sign a separate consent form for the surgery. Additional routine blood tests (about 2 tablespoons) and a PET scan will be done before surgery.

If you have tumors removed, around 28 days after the surgery, you will be given 8 additional cycles of bevacizumab given the same way as before surgery.

Around 4-6 weeks after the final chemotherapy treatment, you will have follow-up CT scans of the abdomen and pelvis, a chest x-ray or CT scan of the chest, and a routine blood test (about 2 tablespoons). These tests will be repeated every 3 months for the first 3 years after surgery, every 6 months for the 4th and 5th year after surgery, and then once a year for the rest of your life. PET scans will be done once a year to check on the status of the disease.

This is an investigational study. Oxaliplatin, 5-FU, leucovorin, and bevacizumab are FDA approved and commercially available for the treatment of this disease. However, their use together in this study is investigational. Up to 42 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have hepatic colorectal metastasis confirmed by percutaneous or intraoperative hepatic tumor biopsy.
2. Patients must have radiological evidence of measurable liver metastasis with helical CT scan (1 cm or greater in greatest transverse dimension).
3. Patients with synchronous disease and resectable intact primary tumors are eligible.
4. Colorectal liver metastases will be determined to be unresectable by a surgeon with expertise in hepatic surgery (equal to or greater than 10 resections performed in a year). A patient is defined as unresectable when distribution and extent of disease preclude margin negative resection (tumor contact with or involvement of all three major hepatic veins or portal confluence or a combination of involvement of main branches of portal veins and hepatic veins), but two adjacent hepatic segments with adequate vascular inflow and outflow are relatively spared (contain 4 or fewer lesions).
5. Performance status: Zubrod 0 or 1.
6. Patients with a prior history of non-colorectal cancer may be included if there is no evidence of malignancy for at least 5 years from last treatment and no evidence of recurrence. In addition, patients with completely resected non-melanoma skin cancer or cervical carcinoma in-situ may be included.
7. Radiological baseline studies shall be completed within 21 days of protocol registration.
8. Laboratory data as follows (within 21 days of protocol registration): Adequate bone marrow as evidenced by; Hemoglobin greater than or equal to 9.0 g %; White blood cell count greater than or equal to 3,000 cells/mm; Platelet count greater than or equal to 100,000 cells/mm(3); Absolute neutrophil count greater than or equal to 1500/mm(3).
9. Continued from inclusion # 9: Laboratory data as follows (within 21 days of protocol registration): Adequate renal function as evidenced by; Creatinine less than or equal to 1.5 mg/dL or estimated creatinine clearance greater than or equal to 60 cc/min; Urinalysis: less than or equal to trace proteinuria. If greater than trace proteinuria exists, a 24- hour urine collection for assessment of protein must demonstrate less than 500 mg of protein/24 hours.
10. Continued from inclusion #10: Laboratory data as follows (within 21 days of protocol registration): Adequate hepatic function as evidenced by; Total Bilirubin less than or equal to 2.0 mg %; Alanine aminotransferase less than or equal to 280 IU/L; Aspartate aminotransferase less than or equal to 230 IU/L; International normalized ratio less than or equal to 2.0.
11. Women must not be pregnant or lactating. Women of childbearing potential must have a negative Beta-HCG serum pregnancy test and to refrain from breast-feeding, as specified in the informed consent given the unknown risk of teratogenicity of agents in the study. Patients of childbearing potential agree to use an effective form of contraception during the study and for 90 days following the last dose of study medication.
12. Age greater than or equal to 18 years.
13. Coumadin, 1 mg, for patency of central venous catheter or therapeutic doses of coumadin (INR less than or equal to 3) permitted.
14. Patients or their legally authorized representative must agree to participate, be able to read, understand and provide informed consent to participate in the trial.
15. Patients must be recovered from both acute and late effects of any prior surgery, radiotherapy or other antineoplastic therapy.

Exclusion Criteria:

1. Patients with surgically resectable colorectal liver metastases.
2. Patients with evidence of unresectable extrahepatic disease.
3. Patients with CNS metastases.
4. Patients with diffusely distributed bilateral hepatic metastases without sparing of two adjacent hepatic segments.
5. Patients who have previously undergone chemotherapy treatment for metastatic disease.
6. Patients who developed metastatic disease less than or equal to 6 months from adjuvant chemotherapy for stage II or stage III colorectal cancer.
7. Patients who have ever received bevacizumab.
8. Previous or concurrent treatment of hepatic metastatic disease with resection, radiotherapy, radiofrequency ablation, cryotherapy/other ablative techniques, or hepatic artery infusion chemotherapy.
9. Patients who underwent a major invasive surgical procedure or open biopsy within 28 days prior to registration.
10. Patients who underwent colonoscopy, core biopsy, or fine needle aspiration within 7 days prior to registration.
11. Patients who had an arterial thromboembolic event, including transient ischemic attack (TIA), cerebrovascular accident (CVA), unstable angina, or myocardial infarction (MI) within 12 months of registration. Patients must not have greater than or equal to Grade 2 peripheral vascular disease.
12. Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, cardiac disease NYHA class III or IV, unstable angina pectoris, unstable cardiac arrhythmia or tachycardia (heart rate greater than or equal to 100 beats per minute), poorly controlled hypertension (systolic blood pressure greater than or equal to 200 mmHg or diastolic blood pressure greater than or equal to 100 mmHg) or psychiatric illness/social situations that would limit compliance with study requirements are excluded.
13. Patients with preexisting chronic hepatic disease (chronic active hepatitis B or C, cirrhosis), which would preclude surgical resection of metastases.
14. Patients with known hypersensitivity to any of the components of oxaliplatin, 5-fluorouracil, leucovorin or bevacizumab (AVASTIN™).
15. Patients who have received chemotherapy within 30 days of the first scheduled day of protocol treatment.
16. Patients who received radiotherapy within 4 weeks of trial entry.
17. Patients who are receiving concurrent investigational therapy or who have received investigational therapy within 30 days of the first scheduled day of protocol treatment (investigational therapy is defined as treatment for which there is currently no regulatory authority approved indication).
18. Peripheral neuropathy greater than or equal to Grade 2.
19. Patients with an active infection or with a fever greater than or equal to 38.5 degrees C within 3 days of the first scheduled day of protocol treatment.
20. Patients with known autoimmune disease including HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2005-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eddie Abdalla, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 11/16/05 through 08/24/07. All participants recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Study terminated early due to slow accrual. Two patients recruited, both were taken off study (one at surgery and the second prior to adjuvant care).
Period: Overall Study
Arm/Group | FOLFOX-B
Started | 2
Completed | 0
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | FOLFOX-B
Number analyzed (Participants) | 2
Age Continuous [Mean (Full Range); unit: years] | 46 [36 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Complete Gross Resection Rate
Description: Complete gross resection rate for patients with initially unresectable hepatic colorectal metastasis who are treated with a combination of oxaliplatin/ 5-fluorouracil/ leucovorin/ bevacizumab (Number of Resectable versus Not Resectable Patients).
Time Frame: Over 4 year study period
Population: Intended analysis was per protocol. Study terminated early, leading to only two (2) patients recruited, one not eligible for study and second inevaluable.
Arm/Group | FOLFOX-B
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 21 Months
Arm/Group | FOLFOX-B
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFOX-B (N=2)
Fever (General disorders) | 1 (1)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 1 (1)
Syncope (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No